CLINICAL TRIAL: NCT00545337
Title: 26-week, International Multicenter, Open, Non-randomized Phase III Clinical Trial for Evaluation of Efficacy and Safety of Insulin Glulisine (HMR1964) Injected Subcutaneously in Subjects With Type 1 Diabetes Mellitus Also Using Insulin Glargine
Brief Title: Glulisine + Lantus in Type I Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3505UA
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insuline glulisine

SUMMARY:
To evaluate the efficacy (in terms of change HbA1c from baseline to endpoint) and safety (in terms of adverse events, clinical chemistry, lipids, hematology) of insulin glulisine (HMR 1964) in subjects with type I diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* type I diabetes mellitus (onset of diabetes under the age of 40),
* an HbA1c range of >6.5 - <11%,
* and on multiple injection regimen (more than 1 year of continuous insulin treatment),
* body mass index <35.

Exclusion Criteria:

* Active proliferative diabetic retinopathy,
* Diabetes other than type I diabetes mellitus,
* Pancreatectomised subjects,
* Subjects who have undergone pancreas and or islet cell transplants,
* Requiring treatment with not permited drugs during the study,
* Previous treatment (in the period not less than 1 month before the beginning of the trial) with insulin glargine,
* Hypersensitivity to insulin,
* Major systemic diseases,
* Impaired hepatic or renal function

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c | from baseline to endpoint

SECONDARY OUTCOMES:
Change of HbA1c | from baseline to week 26
Blood glucose parameters, hypoglycemic episodes and dosage of the mealtime and basal insulins | from baseline to endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Volodymyr Moshchych, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Kiev, Ukraine